CLINICAL TRIAL: NCT03584893
Title: An Observational Study With Retrospective and Prospective Evaluations to Determine the Prevalence of Cerebrotendinous Xanthomatosis (CTX) Disorder in Juvenile Cataract Cases in Turkey
Brief Title: The Prevalence of CTX Disorder in Juvenile Cataract Cases in Turkey
Acronym: GEN-EYE-I
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: TRPHARM (Industry)
Collaborators: Klinar CRO (Other); Düzen Laboratories Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: TR-CTX-001
Record Dates: First submitted 2018-06-19; First posted 2018-07-12 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Cerebrotendinous Xanthomatosis
Keywords: Juvenile Cataract; CTX; Diarrhea; Neonatal Jaundice; Xanthoma
MeSH Terms: conditions — Xanthomatosis, Cerebrotendinous; Diarrhea; Jaundice, Neonatal; Xanthomatosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood samples will be sent to Duzen Laboratories in Ankara and analyzed for cholestanol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Epidemiologic observational study cohort: All patients over 1 year old diagnosed as idiopathic bilateral juvenile cataracts will be included in the study at the study sites.
  Interventions: Procedure: Blood sampling for Cholestanol Analysis

INTERVENTIONS:
Procedure: Blood sampling for Cholestanol Analysis — Cholestanol analysis will be performed to see the Rate of juvenile cataract patients whose cholestanol test result is above threshold (3.75 mg/mL) and suspected CTX cases

SUMMARY:
Epidemiologic observational study. Study will include two phases:

1. Retrospective cross-sectional phase: At this stage of the study, retrospective screenings are carried out at study sites and all juvenile cataract cases are planned to be determined.
2. Prospective phase: At this stage of the study, identified juvenile cataract cases as a result of retrospective screenings will be called to be invited to the sites and blood samples will be obtained for the cholestanol tests for the cases that have given Informed Consent.

This observational study is designed in two phases; retrospective and prospective. Retrospective part includes screening the patient database and / or patient files at ophthalmology clinics participating in the study and identifying patients diagnosed with idiopathic juvenile cataracts. The data of patients with idiopathic juvenile cataracts will be reviewed and the data of the patients meeting the inclusion/exclusion criteria will be recorded. Once this phase is completed, the prospective phase of the study will start and the patients meeting the criteria will be invited to the site to participate in the study. Current data will be collected from the patients who agree to participate in the study and the clinical status of the patients will be evaluated according to the Mignarri index. In addition, blood will be obtained from all patients to diagnose CTX disease. Blood samples will be sent to Duzen Laboratories in Ankara and analyzed for cholestanol.

ELIGIBILITY:
Inclusion Criteria:

* Providing the written informed consent form
* The patient should be diagnosed with idiopathic bilateral juvenile cataract
* Idiopathic bilateral juvenile cataract should be diagnosed while the patient must be take a day from one year (age)
* Syria ciziten who take their citizenship of Turkey could be enrolled to the study after signing of Informed Consent Form that translated to mother tongue by sworn translation office approved by ethic committee.

Exclusion Criteria:

* If the patient has been diagnosed with CTX before his/her enrollment in the study,
* If the patient has been diagnosed with cataract due to any known reasons other than CTX including cataracts related to trauma,
* If the patient has been diagnosed with cataract due to cataractogenic treatments,
* If the patient has participated in an interventional clinical study within the last 30 days,
* If the patient and/or his/her legal representative does not provide consent to participate in the study,
* If the patient will not be able to fulfill study requirements according to the investigator's opinion,
* If the patient had used cholic acid or chenodeoxycholic acid on or before the date of participation in the study
* Pregnancy and/or lactation
* Syria citizen that have not Turkey citizenship will not enroll to the study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients over 1 year old diagnosed as idiopathic bilateral juvenile cataracts will be included in the study at the study sites.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of juvenile cataract patients | "through study completion, an average of 3 years"
  Rate of juvenile cataract patients whose cholestanol test result is above threshold (3.75 mg/mL) and suspected CTX cases

SECONDARY OUTCOMES:
CTX history in family | "through study completion, an average of 3 years"
  The history of the disease will be assessed from the patient records and by interview
Presence of consanguineous marriage | "through study completion, an average of 3 years"
  Presence of consanguineous marriage
The frequency of the systemic findings | "through study completion, an average of 3 years"
  The frequency of the following systemic findings:
  * Tendon xanthomas
  * Chronic diarrhea
  * Prolonged neonatal jaundice
  * Early osteoporosis
The frequency of the neurological symptoms | "through study completion, an average of 3 years"
  The frequency of the following neurological symptoms:
  * Cerebellar ataxia
  * Spastic paraparesis
  * Disruption of dentate nucleus signal detected by MRI
  * Intellectual disability
  * Psychiatric disorders
  * Epilepsy
  * Parkinson
  * Polyneuropathy

CONTACTS AND LOCATIONS:
Locations (36):
- Turkey (Türkiye) (36):
  - Adana Başkent University School of Medicine, Adana
  - Adana State Hospital, Adana
  - Çukurova University Medical Faculty Department of Ophtalmology, Adana
  - Ankara Training and Research Hospital, Ankara
  - Ankara University Medical Faculty Department of Ophtalmology, Ankara
  - Başkent University School of Medicine, Ankara
  - Dünya Göz Hospital, Ankara
  - Hacettepe University Medical Faculty Department of Ophtalmology, Ankara
  - Health Sciences University Ankara State Hospital, Ankara
  - SBU Gülhane Training and Research Hospital, Ankara
  - Ulucanlar Göz Training Hospital, Ankara
  - Akdeniz University Medical Faculty Department of Ophtalmology, Antalya
  - Bursa Yüksek İhtisas Training and Research Hospital, Bursa
  - Uludağ University Medical Faculty Department of Ophtalmology, Bursa
  - Dicle University School of Medicine, Diyarbakır
  - Fırat University School of Medicine, Elâzığ
  - Osmangazi University Medical Faculty Department of Ophtalmology, Eskişehir
  - Gaziantep University Şahinbey Training and Research Hospital, Gaziantep
  - Istanbul University Istanbul Medical Faculty Department of Ophtalmology, Istanbul
  - İstanbul Haseki Training and Research Hospital, Istanbul
  - İstanbul Health Sciences University Kanuni Sultan Süleyman Training and Research Hospital, Istanbul
  - Marmara University Medical Faculty Department of Ophtalmology, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Prof.Dr.N.Reşat Belger Beyoğlu Göz Training and Research Hospital, Istanbul
  - Dokuz Eylül University Medical Faculty Department of Ophtalmology, Izmir
  - Ege University Medical Faculty Department of Ophtalmology, Izmir
  - İzmir Dr. Behcet Uz Child Diseases and Surgery Training and Research Hospital, Izmir
  - Kayseri Training and Research Hospital, Kayseri
  - Kocaeli University School of medicine, Kocaeli
  - İnönü University School of Medicine, Malatya
  - Mersin University Medical Faculty Department of Ophtalmology, Mersin
  - Sakarya University School of Medicine, Sakarya
  - Ondokuz Mayıs University School of Medicine, Samsun
  - Harran University Research and Application Hospital, Sanliurfa
  - Karadeniz Technical University School of Medicine, Trabzon
  - Van 100. Yıl University Dursun Odabaş Medical Center, Van

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clayton PT (2016) Disorders of Bile Acid Synthesis. In: Saudubray JM, Baumgartner MR, Walter J (eds) Inborn metabolic diseases: diagnosis and treatment, 6th ed. Springer-Verlag, Heidelberg, pp 465- 477
- [Background] Nie S, Chen G, Cao X, Zhang Y. Cerebrotendinous xanthomatosis: a comprehensive review of pathogenesis, clinical manifestations, diagnosis, and management. Orphanet J Rare Dis. 2014 Nov 26;9:179. doi: 10.1186/s13023-014-0179-4. PMID 25424010
- [Background] Federico A, Dotti MT, Gallus GN (2003) Cerebrotendinous Xanthomatosis. In: Pagon RA, Adam MP, Ardinger HH, et al. (eds) GeneReviews Seattle (WA): University of Washington, Seattle, 1993- 2017 (updated 2016 Apr 14)
- [Background] Fraidakis MJ. Psychiatric manifestations in cerebrotendinous xanthomatosis. Transl Psychiatry. 2013 Sep 3;3(9):e302. doi: 10.1038/tp.2013.76. PMID 24002088
- [Background] Cruysberg JR, Wevers RA, Tolboom JJ. Juvenile cataract associated with chronic diarrhea in pediatric cerebrotendinous xanthomatosis. Am J Ophthalmol. 1991 Nov 15;112(5):606-7. doi: 10.1016/s0002-9394(14)76874-6. No abstract available. PMID 1951610
- [Background] Mignarri A, Gallus GN, Dotti MT, Federico A. A suspicion index for early diagnosis and treatment of cerebrotendinous xanthomatosis. J Inherit Metab Dis. 2014 May;37(3):421-9. doi: 10.1007/s10545-013-9674-3. Epub 2014 Jan 18. PMID 24442603
- [Background] Verrips A, Hoefsloot LH, Steenbergen GC, Theelen JP, Wevers RA, Gabreels FJ, van Engelen BG, van den Heuvel LP. Clinical and molecular genetic characteristics of patients with cerebrotendinous xanthomatosis. Brain. 2000 May;123 ( Pt 5):908-19. doi: 10.1093/brain/123.5.908. PMID 10775536
- [Background] Salen G, Steiner RD. Epidemiology, diagnosis, and treatment of cerebrotendinous xanthomatosis (CTX). J Inherit Metab Dis. 2017 Nov;40(6):771-781. doi: 10.1007/s10545-017-0093-8. Epub 2017 Oct 4. PMID 28980151
- [Background] Cali JJ, Hsieh CL, Francke U, Russell DW. Mutations in the bile acid biosynthetic enzyme sterol 27-hydroxylase underlie cerebrotendinous xanthomatosis. J Biol Chem. 1991 Apr 25;266(12):7779-83. PMID 2019602
- [Background] Yahalom G, Tsabari R, Molshatzki N, Ephraty L, Cohen H, Hassin-Baer S. Neurological outcome in cerebrotendinous xanthomatosis treated with chenodeoxycholic acid: early versus late diagnosis. Clin Neuropharmacol. 2013 May-Jun;36(3):78-83. doi: 10.1097/WNF.0b013e318288076a. PMID 23673909
- [Background] Khan AO, Aldahmesh MA, Mohamed JY, Alkuraya FS. Juvenile cataract morphology in 3 siblings not yet diagnosed with cerebrotendinous xanthomatosis. Ophthalmology. 2013 May;120(5):956-60. doi: 10.1016/j.ophtha.2012.10.032. Epub 2013 Jan 31. PMID 23375591